CLINICAL TRIAL: NCT02343458
Title: A Randomized, Double-Blind, Chronic Dosing (24 Weeks), Placebo-Controlled, Parallel Group, Multi-Center Study to Assess the Efficacy and Safety of PT003, PT005, and PT001 in Subjects With Moderate to Very Severe COPD, Compared With Placebo
Brief Title: Study to Assess the Efficacy and Safety of PT003, PT005, and PT001 in Subjects With Moderate to Very Severe COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT003014
Record Dates: First submitted 2015-01-06; First posted 2015-01-22 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GFF MDI (PT003) (Experimental): Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI; PT003); Glycopyrronium and Formoterol Fumarate Inhalation Aerosol administered as 2 inhalations twice-daily (BID)
  Interventions: Drug: GFF MDI (PT003)
- FF MDI (PT005) (Experimental): Formoterol Fumarate Metered Dose Inhaler (FF MDI; PT005); Formoterol Fumarate Inhalation Aerosol administered as 2 inhalations twice-daily (BID)
  Interventions: Drug: FF MDI (PT005)
- GP MDI (PT001) (Experimental): Glycopyrronium Metered Dose Inhaler (GP MDI; PT001); Glycopyrronium Inhalation Aerosol administered as 2 inhalations twice-daily (BID)
  Interventions: Drug: GP MDI (PT001)
- Placebo MDI (Placebo Comparator): Placebo (matching) for GFF MDI, FF MDI, and GP MDI administered as 2 inhalations twice-daily (BID)
  Interventions: Drug: Placebo MDI

INTERVENTIONS:
Drug: GFF MDI (PT003) — Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI; PT003); Glycopyrronium and Formoterol Fumarate Inhalation Aerosol administered as 2 inhalations twice-daily (BID)
  Other Names: Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI; PT003); Glycopyrronium and Formoterol Fumarate Inhalation Aerosol
  Arms: GFF MDI (PT003)
Drug: FF MDI (PT005) — Formoterol Fumarate Metered Dose Inhaler (FF MDI; PT005); Formoterol Fumarate Inhalation Aerosol administered as 2 inhalations twice-daily (BID)
  Other Names: Formoterol Fumarate Metered Dose Inhaler (FF MDI; PT005); Formoterol Fumarate Inhalation Aerosol
  Arms: FF MDI (PT005)
Drug: GP MDI (PT001) — Glycopyrronium Metered Dose Inhaler (GP MDI; PT001); Glycopyrronium Inhalation Aerosol administered as 2 inhalations twice-daily (BID)
  Other Names: Glycopyrronium Metered Dose Inhaler (GP MDI; PT001); Glycopyrronium Inhalation Aerosol
  Arms: GP MDI (PT001)
Drug: Placebo MDI — Placebo (matching) for GFF MDI, FF MDI, and GP MDI administered as 2 inhalations twice-daily (BID)
  Other Names: Placebo (matching) for GFF MDI, FF MDI, and GP MDI
  Arms: Placebo MDI

SUMMARY:
A chronic dosing (24 weeks) study to assess the efficacy and safety GFF MDI; PT003), FF MDI; PT005, and GP MDI; PT001) in subjects with moderate to very severe COPD, compared with placebo.

DETAILED DESCRIPTION:
A randomized, double-blind, chronic dosing (24 weeks), placebo-controlled, parallel group, multi-center study to assess the efficacy and safety of glycopyrronium and formoterol fumarate inhalation aerosol (GFF; PT003), formoterol fumarate inhalation aerosol (FF; PT005), and glycopyrronium inhalation aerosol (GP; PT001) in subjects with moderate to very severe COPD, compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Non-child bearing potential (ie, physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal); or Child bearing potential, has a negative serum pregnancy test at Visit 1, and agrees to acceptable contraceptive methods used consistently and correctly for the duration of the study.
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS).
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking.
* Forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) ratio of <0.70.
* FEV1 must be <80% predicted normal value calculated using the Third National Health and Nutrition Examination Survey (NHANES III) reference equations. (Or reference norms applicable to other regions).

Exclusion Criteria:

* Significant diseases other than COPD, ie, disease or condition which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study.
* Women who are pregnant or lactating or women of childbearing potential who are not using an acceptable method of contraception.
* Subjects, who in the opinion of the Investigator, have a current diagnosis of asthma.
* Subjects who have been hospitalized due to poorly controlled COPD within 3 months prior to Visit 1 (Screening) or during the Screening Period (Visit 1 to Visit 4).
* Subjects who have poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to Visit 1 (Screening) or during the Screening Period (Visit 1 to Visit 4).
* Subjects with a diagnosis of angle closure glaucoma will be excluded, regardless of whether or not they have been treated. Subjects with a diagnosis of open angle glaucoma who have intraocular pressure controlled with medication(s) are eligible.
* Subjects who have a history of hypersensitivity to β2-agonists, glycopyrronium or other muscarinic anticholinergics, or any component of the MDI.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1756 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, MD, Study Chair — Pearl Therapeutics, Inc.
Locations (135):
- United States (40):
  - Research Site, Andalusia, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Foley, Alabama
  - Research Site, Jasper, Alabama
  - Research Site, Anaheim, California
  - Research Site, Boulder, Colorado
  - Research Site, Clearwater, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Miami, Florida
  - Research Site, Panama City, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Blue Ridge, Georgia
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Edina, Minnesota
  - Research Site, Fridley, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Woodbury, Minnesota
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Gastonia, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Easley, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Seneca, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Johnson City, Tennessee
  - Research Site, Abingdon, Virginia
- China (23):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hefei
  - Research Site, Heshan
  - Research Site, Hohhot
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shengyang
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wuxi
  - Research Site, Xiamen
  - Research Site, Xining
- Czechia (4):
  - Research Site, Jindřichův Hradec
  - Research Site, Ostrava-Hrabuvka
  - Research Site, Prague
  - Research Site, Teplice
- Germany (7):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Grosshansdof
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Wiesbaden
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Gödöllő
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Siófok
  - Research Site, Szeged
- Japan (29):
  - Research Site, Ako-shi
  - Research Site, Asahikawa-shi
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hamamatsu
  - Research Site, Himeji-shi
  - Research Site, Hitachi-Naka
  - Research Site, Itabashi-ku
  - Research Site, Kakogawa-shi
  - Research Site, Kamogawa-shi
  - Research Site, Kanazawa
  - Research Site, Kishiwada-shi
  - Research Site, Kobe
  - Research Site, Koga-shi
  - Research Site, Matsumoto-shi
  - Research Site, Mito
  - Research Site, Nagaoka-shi
  - Research Site, Nagoya
  - Research Site, Naka-gun
  - Research Site, Ohota-ku
  - Research Site, Ōita
  - Research Site, Saiki-shi
  - Research Site, Sendai
  - Research Site, Seto-shi
  - Research Site, Shimotsuga-gun
  - Research Site, Takamatsu
  - Research Site, Toon-shi
  - Research Site, Yanagawa-shi
  - Research Site, Yokohama
- Poland (11):
  - Research Site, Bialystok
  - Research Site, Elblag
  - Research Site, Inowrocław
  - Research Site, Lodz
  - Research Site, Piekary Śląskie
  - Research Site, Rzeszów
  - Research Site, Skierniewice
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Warszawa Targowek
- Russia (4):
  - Research Site, Gatchina
  - Research Site, Moscow
  - Research Site, Pytigorsk
  - Research Site, Saint Petersburg
- South Korea (4):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Seoul
  - Research Site, Wŏnju
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- United Kingdom (4):
  - Research Site, Dundee
  - Research Site, London
  - Research Site, Northwood
  - Research Site, Sidcup

IPD SHARING:
Plan to Share IPD: Yes
AstraZeneca's policy is to share data with researchers if the request is in scope of our policy. The policy and additional information can be found on astrazenecaclinicaltrials.com.

REFERENCES:
- [Derived] Singh D, Hurst JR, Martinez FJ, Rabe KF, Bafadhel M, Jenkins M, Salazar D, Dorinsky P, Darken P. Predictive modeling of COPD exacerbation rates using baseline risk factors. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221107314. doi: 10.1177/17534666221107314. PMID 35815359
- [Derived] Martinez FJ, Lipworth BJ, Rabe KF, Collier DJ, Ferguson GT, Sethi S, Feldman GJ, O'Brien G, Jenkins M, Reisner C. Benefits of glycopyrrolate/formoterol fumarate metered dose inhaler (GFF MDI) in improving lung function and reducing exacerbations in patients with moderate-to-very severe COPD: a pooled analysis of the PINNACLE studies. Respir Res. 2020 May 25;21(1):128. doi: 10.1186/s12931-020-01388-y. PMID 32450869
- [Derived] Martinez FJ, Rabe KF, Lipworth BJ, Arora S, Jenkins M, Martin UJ, Reisner C. Glycopyrrolate/Formoterol Fumarate Metered Dose Inhaler Improves Lung Function versus Monotherapies in GOLD Category A Patients with COPD: Pooled Data from the Phase III PINNACLE Studies. Int J Chron Obstruct Pulmon Dis. 2020 Jan 9;15:99-106. doi: 10.2147/COPD.S229794. eCollection 2020. PMID 32021148
- [Derived] Chen R, Zhong N, Wang HY, Zhao L, Mei X, Qin Z, Huang J, Assam PN, Maes A, Siddiqui S, Martin UJ, Reisner C. Efficacy And Safety Of Glycopyrrolate/Formoterol Fumarate Metered Dose Inhaler (GFF MDI) Formulated Using Co-Suspension Delivery Technology In Chinese Patients With COPD. Int J Chron Obstruct Pulmon Dis. 2020 Jan 8;15:43-56. doi: 10.2147/COPD.S223638. eCollection 2020. PMID 32021143
- See also: Updated cover page — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4150&filename=PT003014%20Statistical%20Analysis%20Plan%2011_01_01%20_Redacted%20updated%2020181003%20PDFA.pdf
- See also: Updated Cover page — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4150&filename=PT003014-05-%20CLINICAL%20STUDY%20PROTOCOL%20Redacted_updated%2020181003%20PDFA.pdf
- See also: Updated Cover page — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4150&filename=PT003014-05-%20CLINICAL%20STUDY%20PROTOCOL%20Redacted%20PDFA.pdf
- See also: Updated cover page — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4150&filename=PT003014%20Statistical%20Analysis%20Plan%20PDFA.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 175 sites in the United States, United Kingdom, Taiwan (TW),South Korea (SK), Russia, Poland, Hungary, Germany, Czech Republic, China, and Japan from April 2015 to August 2017. The entire study period was scheduled to take approximately 30 weeks for each individual subject from the time of screening.
Pre-assignment Details: Subjects were randomized in a 7:6:6:3 scheme (GFF MDI, FF MDI, GP MDI, and Placebo MDI). Randomization was stratified by reversibility to Ventolin HFA and COPD disease severity (moderate vs severe or very severe) to ensure a similar distribution of treatment arms across stratum.
Groups:
- GFF MDI 14.4/9.6 ug: Glycopyrronium, Formoterol Fumarate, Metered Dose Inhalation 14.4/9.6 ug
- FF MDI 9.6 ug: Formoterol Fumarate, Metered Dose Inhalation 9.6 ug
- GP MDI 14.4 ug: Glycopyrronium 14.4 ug Metered Dose Inhalation
- Placebo MDI: Placebo Metered Dose Inhalation
Period: Overall Study
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Started | 555 | 483 | 480 | 238
Completed (1 subject has been captured in CSR who completed the study but had no follow up phone call.) | 494 | 417 | 417 | 200
Not Completed | 61 | 66 | 63 | 38
Not completed — Adverse Event | 15 | 14 | 15 | 3
Not completed — Lack of Efficacy | 3 | 8 | 4 | 8
Not completed — Withdrawal by Subject | 18 | 17 | 23 | 14
Not completed — Physician Decision | 1 | 4 | 2 | 2
Not completed — Lost to Follow-up | 5 | 5 | 3 | 1
Not completed — Protocol Violation | 2 | 5 | 2 | 2
Not completed — Protocol Specified Criteria | 17 | 13 | 14 | 8

BASELINE CHARACTERISTICS:
Population: The data reported from one site was not included in the final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI | Total
Number analyzed (Participants) | 551 | 480 | 474 | 235 | 1740
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: ITT Population
  Years | 64.7 (7.4) | 64.1 (7.6) | 64.0 (8.1) | 63.9 (7.5) | 64.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The data reported from one site was not included in the final analysis
  Participants
    Female | 143 | 115 | 128 | 64 | 450
    Male | 408 | 365 | 346 | 171 | 1290
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
    Asian | 223 | 204 | 181 | 92 | 700
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 12 | 16 | 18 | 6 | 52
    White | 315 | 260 | 275 | 137 | 987
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 at Week 24 of Treatment (US/China Approach)
Description: For the US/China approach, the primary endpoint was the change from baseline in morning pre-dose trough FEV1 at Week 24 of treatment
Time Frame: at week 24
Population: ITT Population - defined as all subjects who were randomized to treatment and received at least 1 dose of the study treatment. Subjects were analyzed according to the treatment they were assigned to at randomization. Number of participants analyzed reflects the ITT population with available data
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 488 | 413 | 412 | 196
mL | 120 [102 to 138] | 47 [28 to 67] | 60 [41 to 80] | -45 [-73 to -17]

2. Primary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 Over Weeks 12-24, Japan Approach
Description: Change from baseline in morning pre-dose trough FEV1 over weeks 12-24, Japan approach
Time Frame: over weeks 12-24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 517 | 436 | 437 | 205
mL | 128 [113 to 143] | 54 [38 to 71] | 74 [58 to 91] | -25 [-49 to -1]

3. Primary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 Over 24 Weeks. Primary Endpoint, EU/SK/TW Approach, Secondary Endpoint US/China Approach.
Description: Change from baseline in morning pre-dose trough FEV1 over 24 weeks. Primary endpoint, EU/SK/TW approach, Secondary endpoint US/China approach.
Time Frame: over 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 541 | 467 | 465 | 225
mL | 135 [121 to 149] | 63 [48 to 78] | 80 [65 to 94] | -20 [-41 to 2]

4. Secondary Outcome: TDI Focal Score Over 24 Weeks, US/China and EU/SK/TW Approach
Description: TDI focal score over 24 Weeks as a Model-Based Average (ITT Population) The TDI is an instrument which measures the changes in the participant's dyspnea from Baseline. The scores in the TDI evaluate ratings for 3 different categories (functional impairment, magnitude of task in exertional capacity, and magnitude of effort). TDI scores ranged from -3 (major deterioration) to +3 (major improvement); total score = -9 to 9
Time Frame: over 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 532 | 458 | 457 | 217
Scores on a scale | 1.6 [1.4 to 1.8] | 1.5 [1.3 to 1.7] | 1.3 [1.1 to 1.5] | 0.8 [0.5 to 1.1]

5. Secondary Outcome: TDI Focal Score Over Weeks 12-24 Japan Approach
Description: TDI focal score over 12-24 Weeks as a Model-Based Average (ITT Population) The TDI is an instrument which measures the changes in the participant's dyspnea from Baseline. The scores in the TDI evaluate ratings for 3 different categories (functional impairment, magnitude of task in exertional capacity, and magnitude of effort). TDI scores ranged from -3 (major deterioration) to +3 (major improvement); total score = -9 to 9
Time Frame: over Weeks 12-24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 515 | 434 | 436 | 205
Scores on a scale | 1.7 [1.5 to 1.9] | 1.5 [1.3 to 1.7] | 1.4 [1.2 to 1.6] | 0.8 [0.5 to 1.1]

6. Secondary Outcome: TDI Focal Score Over 24 Weeks - US/China and EU/SK/TW Approaches -Symptomatic Population
Description: as for outcome 4
Time Frame: over 24 Weeks
Population: Symptomatic Population was defined as all subjects in the ITT Population with CAT scores of ≥15 at Visit 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 244 | 217 | 228 | 108
Scores on a scale | 1.5 [1.2 to 1.7] | 1.3 [1.0 to 1.6] | 1.1 [0.8 to 1.3] | 0.7 [0.3 to 1.2]

7. Secondary Outcome: TDI Focal Score Over Weeks 12-24 - Japan Approach - Symptomatic Population
Description: as for outcome 5
Time Frame: over weeks 12-24
Population: Symptomatic Population was defined as all subjects in the ITT Population with CAT scores of ≥15 at Visit 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 237 | 200 | 218 | 97
Scores on a scale | 1.5 [1.2 to 1.8] | 1.4 [1.0 to 1.7] | 1.1 [0.8 to 1.4] | 0.7 [0.2 to 1.2]

8. Secondary Outcome: Peak Change From Baseline in FEV1 Within 2 Hours Post-dosing at Week 24 US/China Approach
Description: Peak change from baseline in FEV1 within 2 hours post-dosing at Week 24 US/China approach
Time Frame: at week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 490 | 413 | 412 | 196
mL | 358 [338 to 378] | 247 [226 to 269] | 214 [192 to 235] | 55 [24 to 87]

9. Secondary Outcome: Peak Change From Baseline in FEV1 Within 2 Hours Post-dosing Over Weeks 12-24 Japan Approach
Description: Peak change from baseline in FEV1 within 2 hours post-dosing over weeks 12-24 Japan approach
Time Frame: over weeks 12-24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 516 | 436 | 436 | 205
mL | 368 [350 to 386] | 255 [236 to 274] | 228 [209 to 248] | 70 [42 to 98]

10. Secondary Outcome: Peak Change From Baseline in FEV1 Within 2 Hours Post-dosing Over 24 Weeks EU/SK/TW Approach
Description: Peak change from baseline in FEV1 within 2 hours post-dosing over 24 weeks EU/SK/TW approach
Time Frame: over 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 550 | 480 | 474 | 235
mL | 375 [360 to 389] | 277 [261 to 293] | 234 [218 to 250] | 82 [58 to 105]

11. Secondary Outcome: Change From Baseline in SGRQ Total Score at Week 24, US/China Approach
Description: Change from baseline in the SGRQ total score. The SGRQ is a disease-specific questionnaire, self-completed by participants, used to evaluate the effect of GFF MDI, FF MDI and GP MDI on health-related quality of life as compared to placebo in subjects with COPD. The scores range from 0 (minimum, best possible health status) to 100 (maximum, worst possible health status). The SGRQ contains 76 items grouped into three domains (symptoms, activity and impacts). Change from Baseline at a particular visit was calculated as the SGRQ total score at that visit minus Baseline. Change from Baseline in total score of -4 units or lower is considered as clinically meaningful improvement in quality of life
Time Frame: at week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 489 | 415 | 412 | 196
Scores on a scale | -5.3 [-6.4 to -4.2] | -5.6 [-6.8 to -4.4] | -3.7 [-4.8 to -2.5] | -0.9 [-2.6 to 0.8]

12. Secondary Outcome: Change From Baseline in SGRQ Total Score Over Weeks 12-24 , Japan & EU/SK/TW Approach
Description: as for outcome 11
Time Frame: over weeks 12-24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 516 | 436 | 436 | 205
Scores on a scale | -5.2 [-6.1 to -4.3] | -5.0 [-5.9 to -4.0] | -3.6 [-4.6 to -2.6] | -1.7 [-3.1 to -0.3]

13. Secondary Outcome: Change From Baseline in SGRQ Total Score at Week 24 in Symptomatic Population, US/China Approach
Description: as for outcome 11
Time Frame: at week 24
Population: Symptomatic Population was defined as all subjects in the ITT Population with CAT scores of ≥15 at Visit 2n
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 220 | 189 | 202 | 92
Scores on a scale | -6.9 [-8.6 to -5.2] | -7.8 [-9.7 to -5.9] | -3.8 [-5.6 to -2.0] | -1.6 [-4.3 to 1.1]

14. Secondary Outcome: Change From Baseline in SGRQ Total Score Over Weeks 12-24, in Symptomatic Population, Japan & EU/SK/TW Approach
Description: as for outcome 11
Time Frame: over weeks 12-24
Population: Symptomatic Population was defined as all subjects in the ITT Population with CAT scores of ≥15 at Visit 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 237 | 200 | 218 | 97
Scores on a scale | -6.9 [-8.4 to -5.4] | -7.3 [-8.9 to -5.6] | -3.9 [-5.5 to -2.4] | -3.1 [-5.4 to -0.8]

15. Secondary Outcome: Change From Baseline in Average Daily Rescue Ventolin Use Over 24 Weeks in RVU Population, All Approaches
Description: Change from baseline in average daily rescue Ventolin use over 24 weeks in RVU population, all approaches
Time Frame: over 24 weeks
Population: RVU Population - defined as Rescue Ventolin User
Measure: Least Squares Mean (95% Confidence Interval); unit: Puffs/day
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 256 | 232 | 225 | 109
Puffs/day | -1.4 [-1.7 to -1.1] | -1.0 [-1.3 to -0.7] | -0.6 [-0.9 to -0.3] | -0.4 [-0.8 to -0.0]

16. Secondary Outcome: FEV1 Measured at 5 Minutes Post-dose on Day 1
Description: Onset of Action as Assessed by FEV1 Day 1 at 5 Minutes Post-Dose. Reported is the FEV1 measured at 5 minutes post-dose on Day 1 as the first time point when the difference from Placebo was statistically significant
Time Frame: Assessed at 5-minutes post dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 464 | 406 | 403 | 197
Liters | 0.202 [0.191 to 0.212] | 0.186 [0.175 to 0.197] | 0.059 [0.048 to 0.070] | 0.022 [0.006 to 0.038]

17. Secondary Outcome: FEV1 Measured at 15 Minutes Post-dose on Day 1
Description: Onset of Action as Assessed by FEV1 Day 1 at 15 Minutes Post-Dose. Reported is the FEV1 measured at 15 minutes post-dose on Day 1 as the first time point when the difference from Placebo was statistically significant
Time Frame: Assessed at 15-minute post dose on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
Number analyzed (Participants) | 530 | 458 | 453 | 229
Liters | 0.241 [0.230 to 0.252] | 0.220 [0.208 to 0.231] | 0.105 [0.093 to 0.117] | 0.033 [0.016 to 0.050]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed consent throughout the four treatment periods of 24 weeks and up to 10 days following the last dose of study drug.
Description: The Safety Population was defined as all subjects who were randomized to treatment regardless and received at least one dose of study treatment. Serious adverse events collected from the time the subject signed consent up to 14 days following the last dose of study drug.
Arm/Group | GFF MDI 14.4/9.6 ug | FF MDI 9.6 ug | GP MDI 14.4 ug | Placebo MDI
All-Cause Mortality (participants affected / at risk) | 1/551 | 1/480 | 1/474 | 1/235
Serious Adverse Events (participants affected / at risk) | 53/551 | 40/480 | 34/474 | 19/235
Other Adverse Events (participants affected / at risk) | 166/551 | 123/480 | 128/474 | 61/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI 14.4/9.6 ug (N=551) | FF MDI 9.6 ug (N=480) | GP MDI 14.4 ug (N=474) | Placebo MDI (N=235)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 13 (13) | 12 (12) | 7 (7)
Pneumonia (Infections and infestations) | 7 (7) | 2 (2) | 3 (3) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Borrelia Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Colitis ischemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorroids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerous fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudoradicular syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes melitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angel closure glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI 14.4/9.6 ug (N=551) | FF MDI 9.6 ug (N=480) | GP MDI 14.4 ug (N=474) | Placebo MDI (N=235)
Viral upper respiratory tract infection (Infections and infestations) | 50 (56) | 46 (52) | 44 (55) | 16 (17)
Upper respiratory tract infection (Infections and infestations) | 37 (44) | 29 (34) | 33 (40) | 20 (24)
Pneumonia (Infections and infestations) | 9 (9) | 5 (5) | 5 (5) | 6 (6)
Bronchitis (Infections and infestations) | 4 (5) | 6 (7) | 8 (8) | 5 (5)
Pharyngitis (Infections and infestations) | 11 (11) | 4 (4) | 3 (3) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 13 (13) | 12 (12) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 8 (8) | 10 (11) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 7 (7) | 6 (8) | 7 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 15 (16) | 5 (5) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT02343458/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT02343458/SAP_001.pdf